CLINICAL TRIAL: NCT06363955
Title: A Randomized Placebo-Controlled Clinical Trial Assessing the Efficacy of a Carbamide Peroxide Mouthwash for Oral Wound Healing, Postoperative Symptoms, Xerostomia Relief, and Oral Hygiene Following Diagnostic Biopsy of Minor Labial Salivary Glands for Sjögren's Syndrome Investigation
Brief Title: Assessing the Efficacy of a Carbamide Peroxide Mouthwash for Oral Wound Healing, Oral Hygiene and Xerostomia Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Ioulia And Irene Tseti Pharmaceutical Laboratories S.A. (Industry)
Responsible Party: Principal Investigator, Nikolaos Nikitakis, Professor and Chair, Department of Oral Medicine and Pathology and Hospital Dentistry, School of Dentistry and Dean, School of Dentistry, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNIMOUTH; 750/13.02.2023 (Other: National and Kapodistrian University of Athens)
Record Dates: First submitted 2024-04-05; First posted 2024-04-12 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Wound Heal; Oral Dryness; Postoperative Pain; Sjogren's Syndrome; Biopsy Wound; Mouth; Wound; Mouth Dryness; Dental Plaque; Gingival Inflammation
Keywords: Oral Wound Healing; Oral Biopsy; Postoperative Symptoms; Oral Hygiene; Mouthwash; Hydrogen Carbamide; Hydrogen Peroxide; Sjogren's Syndrome; Minor Salivary Glands Biopsy; Primary Intention Healing; Dental Plaque; Gingival Inflammation
MeSH Terms: conditions — Xerostomia; Pain, Postoperative; Sjogren's Syndrome; Wounds and Injuries; Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: This trial is designed as a prospective, randomized, placebo-controlled, triple blinded, with two parallel groups and an equal allocation ratio in all groups. In this study, the intervention consists of delivery of a hydrogen carbamide/peroxide mouthwash or placebo mouthwash, made by the same manufacturer.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbamide Peroxide Mouthwash (Experimental): A mouthwash containing carbamide proxide/hydrogen peroxide as active ingredient
  Interventions: Device: Carbamide Peroxide Mouthwash
- Placebo (Placebo Comparator): A mouthwash that looks, smells and tastes like the experinmental mouthwash without active ingredients
  Interventions: Device: Placebo mouthwash

INTERVENTIONS:
Device: Carbamide Peroxide Mouthwash — The experinmental mouthwah is a solution containing 4.3% w/v hydrogen carbamide, which breaks down to 1.51% w/v hydrogen peroxide, serving as the active ingredient. Participants rinse (swish and spit) with the mouthwash three times a day for one minute each time, using a 10ml quantity (as indicated by a marking line inside the bottle cap) for a total of 14 days, starting from day 0, i.e. the day of the biopsy (see procedure in the detailed description). Consumption of liquid or solid foods should be avoided for at least thirty minutes following each rinse. Participants are asked to maintain their usual oral hygiene routine. It is a Class IIa, CE-marked medical device made and distributed by Intermed S.A. and Ioulia And Irene Tseti Pharmaceutical Laboratories S.A.
  Other Names: Hydrogen Peroxide Mouthwash
  Arms: Carbamide Peroxide Mouthwash
Device: Placebo mouthwash — Placebo mouthwash is a similar (look-and-taste-alike) solution to the experinmental mouthwash made by the same manufacturer, without active ingredients. Participants rinse (swish and spit) with the mouthwash three times a day for one minute each time, using a 10ml quantity (as indicated by a marking line inside the bottle cap) for a total of 14 days, starting from day 0, i.e. the day of the biopsy (see procedure in the detailed description). Consumption of liquid or solid foods should be avoided for at least thirty minutes following each rinse. Participants are asked to maintain their usual oral hygiene routine.
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of a carbamide peroxide mouthwash regarding oral wound healing, postoperative symptoms, xerostomia (dry mouth) and oral hygiene improvement. Study participants have reported dry mouth and are scheduled for a diagnostic biopsy of minor labial salivary glands to investigate Sjögren's Syndrome, following consultation with their rheumatologist. This is a standardized diagnostic procedure that leads to healing by primary intention (i.e. wound edges are closely re-approximated with sutures).

Researchers are comparing this mouthwash with a placebo (a look-and-taste-alike substance that contains no active ingredients) to see if it is helpful with healing of wounds in the mouth and associated symptoms, improving dry mouth and/or oral hygiene. Carbamide peroxide breaks down to hydrogen peroxide and urea and shows antiseptic and antimicrobial properties and it might help with the parameters to be assessed. Participants randomly get the carbamide peroxide mouthwash or the placebo one to use for 14 days after the biopsy. The investigators will not know which one they are providing as the bottles will be identical.

Oral wound healing, postoperative symptoms (such as pain, eating and speech difficulties), oral hygiene (dental plaque and gingival inflammation), improvement of dry mouth and quality of life are assessed during a 14-day period after the biopsy. Participants are required to visit the clinic three times, one for the initial consultation and the biopsy, one at 7 days and one at 14 days after the biopsy. They are asked to fill in some questionnaires, while certain procedures (such as measuring saliva) and assessments (like evaluating the dental plaque and gingival inflammation) take place. During the first week they, also, keep a diary of their symptoms, as instructed.

DETAILED DESCRIPTION:
This is a prospective, randomized, triple-blind, placebo-controlled clinical trial and post-market clinical follow-up (PMCF) study, expected to last approximately 12 months. All procedures/visits/examinations are taking place in the Oral Medicine and Pathology Clinic at the School of Dentistry, National and Kapodistrian University of Athens, Greece. Participants with reported dry mouth are scheduled for a diagnostic biopsy of minor labial salivary glands to investigate Sjögren's Syndrome, following consultation with their rheumatologist. This is a standardized diagnostic procedure that leads to healing by primary intention. After checking if they comply with the study's criteria, they are informed about the study and the biopsy procedure (including possible complications) and they sign the Ιnformed Consent Form.

All biopsies are obtained from the lower lip with a 12 - 15 mm linear incision. After blunt dissection of the borders, 5-7 lobules of minor salivary glands are removed by dissection with the scalpel or a curved mosquito forceps and the use of tweezers. Attention is paid not to injure nerve branches or vessels. Adequate hemostasis is achieved by manual pressure, and the incision is closed by simple interrupted non-absorbable 4/0 silk sutures at equal distances. Participants are instructed to have cold, soft diet for the day and use ice packs externally for 1-2 hours after the procedure. Use of 500mg paracetamol up to 3 times is permitted for day 0. Following their normal oral hygiene routine (brushing and toothpaste) is suggested.

Subsequently, they are assigned randomly in a 1:1 ratio to receive either a carbamide peroxide mouthwash or a placebo comparator, i.e. a look-alike substance that lacks active ingredients. Both participants and investigators are masked. Follow-up examinations are conducted at 7 and 14 days. On day 7 the sutures are cut.

The evaluation includes:

• oral wound healing (primary intention) assessed by scores (primary outcome)

and secondarily:

* oral wound healing via measuring the incision/wound length
* postoperative symptoms (such as pain, eating and speech difficulties)
* quality of life assessed by a questionnaire
* improvement of dry mouth through subjective and objective measurements
* oral hygiene via plaque and gingival indices.

All data are anonymized and the outcome assessors are masked.

The mouthwash used in the experinmental/test group is a Class IIa, CE-marked (Conformité Européenne) medical device. This mouthwash contains hydrogen carbamide that breaks down to hydrogen peroxide and urea. Hydrogen peroxide has antiseptic and antimicrobial properties, as well the ability to mechanically clean affected areas by producing an oxygenated foam, while urea shares antiseptic and antimicrobial abilities as well and can enhance the pH of the oral cavity. These substances have been used in wound healing either in skin or intraorally, as well as in oral hygiene for a long time. However, to date, no clinical trial examining the use of a hydrogen carbamide/peroxide product in oral wound healing, postoperative symptoms or dry mouth has been reported. Published clinical studies on the control of dental plaque and periodontal inflammation exhibit partially conflicting results.

ELIGIBILITY:
Inclusion criteria

1. Age >18 years
2. Patients requiring lower lip salivary gland biopsy for investigation of Sjögren's syndrome
3. Patients with subjective dry mouth, i.e. who have recorded ≥30mm in at least one of the first 4 questions of the VAS (Visual Analogue Scale) questionnaire according to Pai et al, 2001
4. Able to use the study products (rinse - swish and spit)
5. Agreeing to abstain from the use of any products for xerostomia other than the products provided by the study.
6. Patients who are legally competent and able to understand the information about the study, have been informed of the nature, scope and utility of the study, voluntarily agree to participate and have signed the consent form.

Exclusion criteria

1. Age <18 years
2. Total number of teeth in the oral cavity <10
3. Existence of orthodontic appliances
4. Current use of bleaching trays
5. Presence or history of oral malignant lesions
6. Existence of viral or other infections of the oral cavity or pathology that could interfere with the primary outcomes of the study (e.g. oral vesicobullous disorders)
7. Currently undergoing and/or has received radiation therapy to the head or neck (including radioactive iodine therapy)
8. Currently receiving or has received within the previous 12 months chemotherapy and/or targeted therapies for any malignancy
9. History of acute myocardial infarction and/or vascular stroke during the last 6 months
10. Patients with poor glycemic control (HbA1c ≥ 7% within the previous 3 months according to American Diabetes Association (ADA) recommendations), uncontrolled type I or II diabetes mellitus or other systemic diseases known to affect oral wound healing
11. Use of antibiotics in the last 1 month prior to biopsy or conditions requiring antibiotic prophylaxis
12. Use of any antimicrobial mouthwash in the last 1 month before the biopsy
13. Concurrent immunocompromised status and/or use of immunosuppressant medications (e.g. corticosteroids) and steroid inhalers or nasal sprays within the last 1 month prior to enrollment
14. Use of sialagogues
15. Heavy smokers (those who smoke greater than or equal to 25 cigarettes per day) and tobacco chewers or users of tobacco pouches
16. Received dental treatment during the period included in the study
17. Malnutrition
18. Alcohol abuse and (illicit) drug use disorders
19. Pregnancy or lactation/nursing/breast feeding
20. Known allergy to any of the ingredients of the study products
21. Inability to provide informed consent
22. Participation in another study of an investigational product or device until the primary endpoint is met
23. Other medical condition that, in the opinion of the investigator, may be causing the patient's non-compliance with the clinical investigation plan or confusion in interpreting the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Assessment of wound healing based on the modified Landry Healing Index on day 14 | Day 14
  Healing will be measured clinically using specific scores. The modified Landry Healing Index consists of the assessment of 5 clinical parameters (tissue color, bleeding on palpation, presence of granulation tissue, presence of suppuration, and healing of the surgical margin). As the initial index referred to gingival healing, it was slightly modified as in other studies, so that it refers to oral mucosal healing. The index values range from 1 to 5, where 1 corresponds to "very poor healing" and 5 to "excellent healing". Comparisons will be made between the carbamide peroxide mouthwash versus the placebo group.
Assessment of wound healing based on a modified version of the Early Wound Healing Score (EHS) on day 14 | Day 14
  Healing will be measured clinically using specific scores. The EHS is composed of 3 parameters: clinical signs of re-epithelization (CSR), clinical signs of haemostasis (CSH), and clinical signs of inflammation (CSI). Zero, 3, 4 or 6 points are used to evaluate CSR (modified by adding point 4), whereas 0, 1, or 2 points are used for CSH and CSI. The EHS is generated by the summation of the points of these 3 parameters. The EHS for ideal wound healing is 10 points, while the worst possible score is 0 points. Comparisons will be made between the carbamide peroxide mouthwash versus the placebo group.
Assessment of wound healing based on the modified Landry Healing Index on day 7 | Day 7
  Healing will be measured clinically using specific scores. The modified Landry Healing Index consists of the assessment of 5 clinical parameters (tissue color, bleeding on palpation, presence of granulation tissue, presence of suppuration, and healing of the surgical margin). As the initial index referred to gingival healing, it was slightly modified as in other studies, so that it refers to oral mucosal healing. The index values range from 1 to 5, where 1 corresponds to "very poor healing" and 5 to "excellent healing". Comparisons will be made between the carbamide peroxide mouthwash versus the placebo group.
Assessment of wound healing based on a modified version of the Early Wound Healing Score (EHS) on day 7 | Day 7
  Healing will be measured clinically using specific scores. The EHS is composed of 3 parameters: clinical signs of re-epithelization (CSR), clinical signs of haemostasis (CSH), and clinical signs of inflammation (CSI). Zero, 3, 4 or 6 points are used to evaluate CSR (modified by adding point 4), whereas 0, 1, or 2 points are used for CSH and CSI. The EHS is generated by the summation of the points of these 3 parameters. The EHS for ideal wound healing is 10 points, while the worst possible score is 0 points. Comparisons will be made between the carbamide peroxide mouthwash versus the placebo group.

SECONDARY OUTCOMES:
Postoperative symptoms (pain, eating and speech difficulty) during the first week (at home) | Days 0, 1, 2, 3, 4, 5 and 6
  Participants will be given a pain diary (PD) to complete at home daily at the end of the day, from day 0 to day 6, with instructions for its completion. Specifically, the participants will record: the greatest intensity of the postoperative pain, as perceived (Numerical and Visual Scale, ranked 0-10), difficulty in eating (Yes/No), difficulty in speaking (Yes/No) and whether any analgesic treatment, apart from the one recommended for day 0, has been necessary (No or Yes: Which one?). Comparisons will be made between the two groups for every day from day 0 to day 6.
Postoperative symptoms (pain, eating and speech difficulty) on day 7 | Day 7
  During the visit in day 7, participants will be asked to record: the greatest intensity of the postoperative pain, as perceived (Numerical and Visual Scale, ranked 0-10), difficulty in eating (Yes/No), difficulty in speaking (Yes/No) and whether any analgesic treatment has been necessary (No or Yes: Which one?). Comparisons will be made between the two groups.
Postoperative symptoms (pain, eating and speech difficulty) on day 14 | Day 14
  During the visit in day 14, participants will be asked to record: the greatest intensity of the postoperative pain, as perceived (Numerical and Visual Scale, 0-10), difficulty in eating (Yes/No), difficulty in speaking (Yes/No) and whether any analgesic treatment has been necessary (No or Yes: Which one?). Comparisons will be made between the two groups.
Wound healing based on the incision/wound length | Days 0, 7 and 14
  The incision/wound length will be measured in milimeters (mm) during every visit using a UNC 15 (North Carolina) periodontal probe. Standardized pictures will be also taken with an angulation perpendicular to the wound. The same periodontal probe will be placed by the wound as a reference scale. Comparisons will be made between the two groups (mean changes from day 7 to 0, day 14 to 0 and day 14 to 7).
Subjective oral dryness symptoms (8-item VAS questionnaire) | Days 0, 7 and 14
  During all the visits, patients complete a 8-item 100 mm Visual Analog Scale (VAS) questionnaire developed by Pai et al, 2001 for subjective scoring xerostomia symptoms, namely: difficulty in speaking due to dryness, difficulty in swallowing due to dryness (0 mm: not difficult at all, 100 mm: very difficult), rating the amount of saliva in the mouth (0 mm: a lot, 100 mm: none), level of dryness in the mouth, the throat, the lips and the tongue (0 mm: not dry at all, 100 mm: very dry) and the level of thirst (0 mm: not thirsty at all, 100 mm: very thirsty). Comparisons will be made for each item of the questionnaire between the two groups by calculating the changes from day 7 to 0, day 14 to 0 and day 14 to 7. Higher values of the changes represent a better outcome.
Observed (objective) signs of oral dryness | Days 0, 7 and 14
  During the clinical exam in each visit, Clinical Oral Dryness Score (CODS) is conducted, which assesses ten key features of dry mouth and allocates one point for each feature. The total score ranges from 0 to 10, with higher scores indicating more severe dry mouth. Comparisons will be made between the two groups on days 7 and 14.
Change in Unstimulated Saliva Flow Rate | Days 0 and 14
  Unstimulated whole saliva is collected in a cap over a 5-minute time period at around the same time of the day on days 0 and 14 and the volume is measured. The Unstimulated Saliva Flow Rate is measured in ml per minute and the change is calculated by subtracting the measurement at day 0 from the measurement at 14 days. Comparisons will be made between the two groups.
Oral Hygiene - Dental Plaque: Full-Mouth Plaque Index | Days 0, 7 and 14
  The Plaque Index (PI) by Silness & Loe 1964 is a score of 0-3 with higher scores indicating greater plaque accumulation. Every tooth is evaluated with a UNC 15 periodontal probe at 4 sites (mesiobuccal, mid-buccal, distobuccal, and lingual) as 0 = No plaque, 1 = A film of plaque adhering to free gingival margin and adjacent area of tooth, which may be seen by using the probe or disclosing solution, 2 = Moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin, which can be seen with the naked eye, 3 = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  The calculation of full mouth index refers to the sum of the measurements on the 4 surfaces of all the teeth examined divided by four and then by the number of teeth examined. The final score ranges from 0-3. Full mouth PI is measured in all visits and comparisons will be made between the two groups on day 7 and 14 (mean changes from baseline).
Oral Hygiene - Gingival Inflammation: Full Mouth Gingival Index | Days 0, 7 and 14
  The Gingival Index (GI) by Loe & Silness 1963 scores from 0 to 3, with higher scores indicating greater inflammation. The examination is performed by sliding the periodontal probe (UNC 15) on the free gums (modification according to Löe - 1967) on all existing teeth of the person. Every tooth is evaluated at 4 surfaces (mesiobuccal, mid-buccal, distobuccal, and lingual). By dividing the sum of the values by 4, the gingival index of the tooth is calculated. The full mouth gingival index is obtained by summing the indices of each tooth divided by the total number of teeth examined. The overall index score, representing inflammation, is rated as mild (mean 0,1-1,0), moderate (1,1-2,0) and severe (2,1-3). Comparisons of the full mouth GI scores will be made between the 2 groups on day 7 and 14 (mean changes from baseline).
Oral Health Related Quality of Life | Day 14
  The Oral Health Impact Profile-14 (OHIP-14) scale is used to measure the participants' oral health related quality of life (OHRQoL) after the procedure. It has seven conceptualized domains (two items per domain - 14 total): functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Participants are asked to rate how frequently they experienced an oral health impact (as described by each item), scoring on a five-point Likert scale: never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4). Thus, OHIP-14 scores can range from 0 to 56. A high total value indicates a high negative impact on the OHRQoL. Comparisons will be made between the two groups on day 14.
Assessment of swelling in the biopsy area | Day 7 and 14
  The existence of swelling in the biopsy area is assessed via a Yes/No question ("Is there swelling in the biopsy area?") during visits on day 7 and 14. Comparisons will be made between the two groups.

OTHER OUTCOMES:
Adverse Events | Day 0, Day 7, Day 14
  Adverse events will be recorded at every visit.
Participant's comments and satisfaction regarding the provided treatment/use of the products | Day 14
  Participants are provided with a 12-item questionnaire to complete during their visit on day 14. Eight of these questions pertain to the improvement in breath odor, taste, gum health, the sensation of mouth cleanliness and freshness, as well as the reduction in gum bleeding, ease of product use, and satisfaction level resulting from product use. These are scored on a four-point Likert scale: 'not at all' (score 1), 'slightly' (score 2), 'very' (score 3), and 'extremely' (score 4). Three questions require a 'Yes' or 'No' response, inquiring whether participants would reuse the product in the event of an oral wound or ulcer, for moisturizing the oral cavity and improving dry mouth, and if they would recommend the product. Lastly, one question addressing compliance will be answered using a four-point Likert scale: 0-2 (score 1), 3-5 (score 2), 6-8 (score 3), and 9+ (score 4). Results will be shown for each group and comparative analyses will be conducted between the two groups.
Compliance | Day 14
  All patients are instructed to return the two initially provided bottles after use to record the remaining quantity. Compliance is further assessed through a question included in the aforementioned questionnaire, specifically addressing missed doses, answered on a four-point Likert scale: 0-2 (score 1), 3-5 (score 2), 6-8 (score 3), and 9+ (score 4).

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Nikitakis, DDS, MD, PhD, Study Chair — School of Dentistry, National and Kapodistrian University of Athens; Nikolaos Apostolidis, DDS, Principal Investigator — School of Dentistry, National and Kapodistrian University of Athens
Locations (1):
- Department of Oral Medicine & Pathology and Hospital Dentistry, School of Dentistry, National and kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
The data that supports the findings of this study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests will be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified investigators whose proposed research has received Institutional Review Board (IRB) approval. Data will be available via a data repository following execution of data use agreement.

REFERENCES:
- [Background] Fox PC. Simplified biopsy technique for labial minor salivary glands. Plast Reconstr Surg. 1985 Apr;75(4):592-3. doi: 10.1097/00006534-198504000-00029. No abstract available. PMID 3983264
- [Background] Marshall MV, Cancro LP, Fischman SL. Hydrogen peroxide: a review of its use in dentistry. J Periodontol. 1995 Sep;66(9):786-96. doi: 10.1902/jop.1995.66.9.786. PMID 7500245
- [Background] Pai S, Ghezzi EM, Ship JA. Development of a Visual Analogue Scale questionnaire for subjective assessment of salivary dysfunction. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Mar;91(3):311-6. doi: 10.1067/moe.2001.111551. PMID 11250628
- [Background] Landry RGTR, Howley T. Effectiveness of benzydamine HCl in the treatment of periodontal post-surgical patients. Res Clinic Forums 1988;10:105-118.
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Osailan SM, Pramanik R, Shirlaw P, Proctor GB, Challacombe SJ. Clinical assessment of oral dryness: development of a scoring system related to salivary flow and mucosal wetness. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Nov;114(5):597-603. doi: 10.1016/j.oooo.2012.05.009. Epub 2012 Sep 7. PMID 22959491
- [Background] Papagiannopoulou V, Oulis CJ, Papaioannou W, Antonogeorgos G, Yfantopoulos J. Validation of a Greek version of the oral health impact profile (OHIP-14) for use among adults. Health Qual Life Outcomes. 2012 Jan 14;10:7. doi: 10.1186/1477-7525-10-7. PMID 22244162
- [Background] Marini L, Rojas MA, Sahrmann P, Aghazada R, Pilloni A. Early Wound Healing Score: a system to evaluate the early healing of periodontal soft tissue wounds. J Periodontal Implant Sci. 2018 Oct 24;48(5):274-283. doi: 10.5051/jpis.2018.48.5.274. eCollection 2018 Oct. PMID 30405935
- [Background] Wennstrom J, Lindhe J. Effect of hydrogen peroxide on developing plaque and gingivitis in man. J Clin Periodontol. 1979 Apr;6(2):115-30. doi: 10.1111/j.1600-051x.1979.tb02190.x. PMID 379049
- [Background] Muniz FWMG, Cavagni J, Langa GPJ, Stewart B, Malheiros Z, Rosing CK. A Systematic Review of the Effect of Oral Rinsing with H2O2 on Clinical and Microbiological Parameters Related to Plaque, Gingivitis, and Microbes. Int J Dent. 2020 Oct 31;2020:8841722. doi: 10.1155/2020/8841722. eCollection 2020. PMID 33178277